CLINICAL TRIAL: NCT00300456
Title: A Multicenter, Randomized, Double-Blind, Prospective Study Comparing the Safety and Efficacy of ABT-335 and Simvastatin Combination Therapy to ABT-335 and Simvastatin Monotherapy in Subjects With Mixed Dyslipidemia
Brief Title: Evaluate Safety and Efficacy of ABT-335 in Combination With Simvastatin in Subjects With Multiple Abnormal Lipid Levels in the Blood
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Maureen Kelly, MD, Abbott
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M05-749
Record Dates: First submitted 2006-03-07; First posted 2006-03-09 (Estimated); Results first posted 2009-03-25 (Estimated); Last update posted 2009-06-03 (Estimated); Status verified 2009-05

CONDITIONS: Dyslipidemia; Coronary Heart Disease; Mixed Dyslipidemia
Keywords: Dyslipidemia; Coronary Heart Disease; Mixed Dyslipidemia
MeSH Terms: conditions — Dyslipidemias; Coronary Disease | interventions — 2-(4-(4-chlorobenzoyl)phenoxy)-2-methylpropanoic acid; Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- A (Active Comparator): ABT-335 + 20 mg simvastatin
  Interventions: Drug: ABT-335; Drug: Simvastatin
- B (Active Comparator): ABT-335 + 40 mg simvastatin
  Interventions: Drug: ABT-335; Drug: Simvastatin
- C (Placebo Comparator): ABT-335 monotherapy
  Interventions: Drug: ABT-335; Drug: Placebo
- D (Placebo Comparator): 20 mg simvastatin monotherapy
  Interventions: Drug: Simvastatin; Drug: Placebo
- E (Placebo Comparator): 40 mg simvastatin monotherapy
  Interventions: Drug: Simvastatin; Drug: Placebo
- F (Placebo Comparator): 80 mg simvastatin monotherapy
  Interventions: Drug: Simvastatin; Drug: Placebo

INTERVENTIONS:
Drug: ABT-335 — 135 mg, daily, 12 weeks
  Arms: A; B; C
Drug: Simvastatin — daily, 12 weeks, see Arm Description for dosage information
  Arms: A; B; D; E; F
Drug: Placebo — Daily, 12 weeks, see Arm Description for placebo information
  Arms: C; D; E; F

SUMMARY:
The purpose of this study is to compare the safety and efficacy of fenofibric acid (ABT-335) + simvastatin combination therapy with ABT-335 and simvastatin monotherapy in subjects with multiple abnormal lipid levels in the blood.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with mixed dyslipidemia
* Subjects agree to utilize adequate birth control methods and to adhere to the American Heart Association (AHA) diet.

Exclusion Criteria:

* Subjects with unstable medical conditions or medical conditions considered inappropriate in a clinical trial.
* Patients who are taking certain medications or unstable dose of specific medications.
* Women who are pregnant or plan on becoming pregnant, or women who are lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 657 (Actual)
Dates: Start 2006-03; Primary Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Global Medical Information, North Chicago, Illinois, United States

REFERENCES:
- [Derived] Bays HE, Roth EM, McKenney JM, Kelly MT, Thakker KM, Setze CM, Obermeyer K, Sleep DJ. The effects of fenofibric acid alone and with statins on the prevalence of metabolic syndrome and its diagnostic components in patients with mixed dyslipidemia. Diabetes Care. 2010 Sep;33(9):2113-6. doi: 10.2337/dc10-0357. Epub 2010 Jun 23. PMID 20573750
- [Derived] Jones PH, Cusi K, Davidson MH, Kelly MT, Setze CM, Thakker K, Sleep DJ, Stolzenbach JC. Efficacy and safety of fenofibric acid co-administered with low- or moderate-dose statin in patients with mixed dyslipidemia and type 2 diabetes mellitus: results of a pooled subgroup analysis from three randomized, controlled, double-blind trials. Am J Cardiovasc Drugs. 2010;10(2):73-84. doi: 10.2165/10061630-000000000-00000. PMID 20136164
- [Derived] Jones PH, Bays HE, Davidson MH, Kelly MT, Buttler SM, Setze CM, Sleep DJ, Stolzenbach JC. Evaluation of a new formulation of fenofibric acid, ABT-335, co-administered with statins : study design and rationale of a phase III clinical programme. Clin Drug Investig. 2008;28(10):625-34. doi: 10.2165/00044011-200828100-00003. PMID 18783301

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Seven subjects were randomized but never treated: 2 were taking a prohibited concomitant medication, 1 did not meet the entry criteria for lipid levels, 1 had an abnormal baseline electrocardiogram, 1 was unable to swallow pills, and 2 withdrew consent.
Groups:
- ABT-335 + 20 mg Simvastatin: ABT-335 + 20 mg simvastatin combination therapy once daily
- ABT-335 + 40 mg Simvastatin: ABT-335 + 40 mg simvastatin combination therapy once daily
- ABT-335: ABT-335 monotherapy once daily
- 20 mg Simvastatin: 20 mg simvastatin monotherapy once daily
- 40 mg Simvastatin: 40 mg simvastatin monotherapy once daily
- 80 mg Simvastatin: 80 mg simvastatin monotherapy once daily
Period: Overall Study
Arm/Group | ABT-335 + 20 mg Simvastatin | ABT-335 + 40 mg Simvastatin | ABT-335 | 20 mg Simvastatin | 40 mg Simvastatin | 80 mg Simvastatin
Started | 119 (For all arms, "started" means treated.) | 118 | 119 | 119 | 116 | 59
Completed | 103 | 102 | 98 | 105 | 99 | 48
Not Completed | 16 | 16 | 21 | 14 | 17 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ABT-335 + 20 mg Simvastatin | ABT-335 + 40 mg Simvastatin | ABT-335 | 20 mg Simvastatin | 40 mg Simvastatin | 80 mg Simvastatin | Total
Number analyzed (Participants) | 119 | 118 | 119 | 119 | 116 | 59 | 650
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 101 | 96 | 98 | 104 | 104 | 48 | 551
  >=65 years | 18 | 22 | 21 | 15 | 12 | 11 | 99
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 57 | 68 | 56 | 61 | 31 | 332
  Male | 60 | 61 | 51 | 63 | 55 | 28 | 318
Region of Enrollment [Number; unit: participants]
  North America | 119 | 118 | 119 | 119 | 116 | 59 | 650

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Change in Triglycerides From Baseline to Final Visit
Description: [(Week 12 triglycerides minus baseline triglycerides)/baseline triglycerides] x 100
Time Frame: Baseline to 12 Weeks (Final Visit)
Population: All randomized subjects with a baseline triglyceride value and at least 1 postbaseline triglyceride value, last observation carried forward
Measure: Mean (Standard Error); unit: percent change
Arm/Group | ABT-335 + 20 mg Simvastatin | ABT-335 + 40 mg Simvastatin | ABT-335 | 20 mg Simvastatin | 40 mg Simvastatin | 80 mg Simvastatin
Number analyzed (Participants) | 113 | 111 | 113 | 116 | 112 | 56
percent change | -37.4 (2.75) | -42.7 (2.77) | -31.7 (2.74) | -14.2 (2.71) | -22.4 (2.76) | -20.2 (3.82)
Statistical Analysis 1: Comparison: ABT-335 + 20 mg Simvastatin vs 20 mg Simvastatin; An n = 92 per arm would provide >99% power to detect a 24% decrease in triglycerides relative to statin monotherapy for each combo therapy dose, assuming an SD of 30%; Test type: Superiority or Other; p < 0.001, ANCOVA — alpha = 0.05, all 3 primary endpoints had to show superiority of combo therapy in order to declare combo therapy successful at a given statin dose, Hochberg method for multiple comparison adjustment for 2 statin doses
Statistical Analysis 2: Comparison: ABT-335 + 40 mg Simvastatin vs 40 mg Simvastatin; An n = 92 per arm would provide >99% power to detect 24% decrease in triglycerides relative to statin monotherapy for each combo therapy dose, assuming an SD of 30%; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]

2. Primary Outcome: Mean Percent Change in High-density Lipoprotein Cholesterol (HDL-C) From Baseline to Final Visit
Description: [(Week 12 HDL-C minus baseline HDL-C)/baseline HDL-C] x 100
Time Frame: Baseline to 12 Weeks (Final Visit)
Population: All randomized subjects with a baseline HDL-C value and at least 1 postbaseline HDL-C value, last observation carried forward
Measure: Mean (Standard Error); unit: percent change
Arm/Group | ABT-335 + 20 mg Simvastatin | ABT-335 + 40 mg Simvastatin | ABT-335 | 20 mg Simvastatin | 40 mg Simvastatin | 80 mg Simvastatin
Number analyzed (Participants) | 105 | 106 | 107 | 114 | 102 | 52
percent change | 17.8 (1.86) | 18.9 (1.86) | 16.2 (1.85) | 7.2 (1.80) | 8.5 (1.89) | 6.8 (2.61)
Statistical Analysis 1: Comparison: ABT-335 + 20 mg Simvastatin vs 20 mg Simvastatin; An n = 92 per arm would provide 98% power to detect a 9% increase in HDL-C relative to statin monotherapy for each combo therapy dose, assuming an SD of 15%; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: ABT-335 + 40 mg Simvastatin vs 40 mg Simvastatin; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]

3. Primary Outcome: Mean Percent Change in Low-density Lipoprotein Cholesterol (LDL-C) From Baseline to Final Visit
Description: [(Week 12 LDL-C minus baseline LDL-C)/baseline LDL-C] x 100
Time Frame: Baseline to 12 Weeks (Final Visit)
Population: All randomized subjects with a baseline LDL-C value and at least 1 postbaseline LDL-C value, last observation carried forward
Measure: Mean (Standard Error); unit: percent change
Arm/Group | ABT-335 + 20 mg Simvastatin | ABT-335 + 40 mg Simvastatin | ABT-335 | 20 mg Simvastatin | 40 mg Simvastatin | 80 mg Simvastatin
Number analyzed (Participants) | 109 | 108 | 107 | 116 | 106 | 55
percent change | -24.0 (1.94) | -25.3 (1.96) | -4.0 (1.96) | -22.4 (1.90) | -31.7 (1.98) | -40.8 (2.69)
Statistical Analysis 1: Comparison: ABT-335 + 20 mg Simvastatin vs ABT-335; An n = 92 per arm would provide >99% power to detect an 11% decrease in LDL-C relative to ABT-335 monotherapy for each combo therapy dose, assuming an SD of 15%; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: ABT-335 + 40 mg Simvastatin vs ABT-335; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]

4. Secondary Outcome: Mean Percent Change in Non-high-density Lipoprotein Cholesterol (Non-HDL-C) From Baseline to Final Visit
Description: [(Week 12 non-HDL-C minus baseline non-HDL-C)/baseline non-HDL-C] x 100
Time Frame: Baseline to 12 Weeks (Final Visit)
Population: All randomized subjects with a baseline non-HDL-C value and at least 1 postbaseline non-HDL-C value, LOCF
Measure: Mean (Standard Error); unit: percent change
Arm/Group | ABT-335 + 20 mg Simvastatin | ABT-335 + 40 mg Simvastatin | ABT-335 | 20 mg Simvastatin | 40 mg Simvastatin | 80 mg Simvastatin
Number analyzed (Participants) | 104 | 104 | 107 | 114 | 103 | 52
percent change | -30.7 (1.48) | -35.0 (1.48) | -17.3 (1.46) | -24.4 (1.43) | -35.9 (1.49) | -40.6 (2.06)

5. Secondary Outcome: Mean Percent Change in Very Low-density Lipoprotein Cholesterol (VLDL-C)From Baseline to Final Visit
Description: [(Week 12 VLDL-C minus baseline VLDL-C)/baseline VLDL-C] x 100
Time Frame: Baseline to 12 Weeks (Final Visit)
Population: All randomized subjects with a baseline VLDL-C value and at least 1 postbaseline VLDL-C value, LOCF
Measure: Mean (Standard Error); unit: percent change
Arm/Group | ABT-335 + 20 mg Simvastatin | ABT-335 + 40 mg Simvastatin | ABT-335 | 20 mg Simvastatin | 40 mg Simvastatin | 80 mg Simvastatin
Number analyzed (Participants) | 109 | 111 | 110 | 112 | 110 | 54
percent change | -38.9 (4.06) | -51.1 (4.03) | -36.9 (4.04) | -19.2 (4.04) | -35.7 (4.06) | -30.0 (5.66)

6. Secondary Outcome: Mean Percent Change in Total Cholesterol From Baseline to Final Visit
Description: [(Week 12 total cholesterol minus baseline total cholesterol)/baseline total cholesterol] x 100
Time Frame: Baseline to 12 Weeks (Final Visit)
Population: All randomized subjects with a baseline total cholesterol value and at least 1 postbaseline total cholesterol value, LOCF
Measure: Mean (Standard Error); unit: percent change
Arm/Group | ABT-335 + 20 mg Simvastatin | ABT-335 + 40 mg Simvastatin | ABT-335 | 20 mg Simvastatin | 40 mg Simvastatin | 80 mg Simvastatin
Number analyzed (Participants) | 112 | 111 | 113 | 116 | 112 | 56
percent change | -23.9 (1.20) | -27.1 (1.21) | -12.4 (1.20) | -19.8 (1.19) | -30.0 (1.21) | -33.6 (1.67)

7. Secondary Outcome: Mean Percent Change in Lipoprotein Apo B (Apo B) From Baseline to Final Visit
Description: [(Week 12 Apo B minus baseline Apo B)/baseline Apo B] x 100
Time Frame: Baseline to 12 Weeks (Final Visit)
Population: All randomized subjects with a baseline ApoB value and at least 1 postbaseline ApoB value, LOCF
Measure: Mean (Standard Error); unit: percent change
Arm/Group | ABT-335 + 20 mg Simvastatin | ABT-335 + 40 mg Simvastatin | ABT-335 | 20 mg Simvastatin | 40 mg Simvastatin | 80 mg Simvastatin
Number analyzed (Participants) | 109 | 110 | 112 | 113 | 112 | 54
percent change | -29.5 (1.47) | -31.2 (1.47) | -17.6 (1.45) | -22.9 (1.45) | -32.7 (1.46) | -38.9 (2.05)

8. Secondary Outcome: Median Percent Change in High-sensitivity C-reactive Protein (hsCRP) From Baseline to Final Visit
Description: [(Week 12 hsCRP minus baseline hsCRP)/baseline hsCRP] x 100
Time Frame: Baseline to 12 Weeks (Final Visit)
Population: All randomized subjects with a baseline hsCRP value and at least 1 postbaseline hsCRP value, LOCF
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | ABT-335 + 20 mg Simvastatin | ABT-335 + 40 mg Simvastatin | ABT-335 | 20 mg Simvastatin | 40 mg Simvastatin | 80 mg Simvastatin
Number analyzed (Participants) | 111 | 110 | 112 | 113 | 112 | 54
percent change | -26.8 (48.27) [-40.9 to 8.2] | -32.1 (48.70) [-51.5 to 9.4] | -15.8 (48.01) [-42.5 to 30.9] | -11.4 (48.18) [-36.0 to 21.4] | -14.8 (48.25) [-40.8 to 11.2] | -19.8 (67.84) [-36.0 to 22.6]

ADVERSE EVENTS:
Arm/Group | ABT-335 + 20 mg Simvastatin | ABT-335 + 40 mg Simvastatin | ABT-335 | 20 mg Simvastatin | 40 mg Simvastatin | 80 mg Simvastatin
Serious Adverse Events (participants affected / at risk) | 1 | 3 | 6 | 1 | 1 | 2
Other Adverse Events (participants affected / at risk) | 65 | 72 | 67 | 60 | 65 | 26
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | ABT-335 + 20 mg Simvastatin | ABT-335 + 40 mg Simvastatin | ABT-335 | 20 mg Simvastatin | 40 mg Simvastatin | 80 mg Simvastatin
Angina pectoris (Cardiac disorders) | 1/119 | 0/118 | 0/119 | 0/119 | 0/116 | 0/59
Angina unstable (Cardiac disorders) | 0/119 | 0/118 | 1/119 | 0/119 | 0/116 | 0/59
Mitral valve incompetence (Cardiac disorders) | 0/119 | 1/118 | 0/119 | 0/119 | 0/116 | 0/59
Myocardial infarction (Cardiac disorders) | 0/119 | 0/118 | 1/119 | 0/119 | 0/116 | 0/59
Colonic polyp (Gastrointestinal disorders) | 0/119 | 0/118 | 0/119 | 1/119 | 0/116 | 0/59
Chest pain (General disorders) | 0/119 | 0/118 | 0/119 | 0/119 | 0/116 | 1/59
Fall (Injury, poisoning and procedural complications) | 0/119 | 0/118 | 1/119 | 0/119 | 0/116 | 0/59
Gun shot wound (Injury, poisoning and procedural complications) | 0/119 | 0/118 | 0/119 | 0/119 | 0/116 | 1/59
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0/119 | 0/118 | 1/119 | 0/119 | 0/116 | 0/59
Cerebrovascular accident (Nervous system disorders) | 0/119 | 1/118 | 0/119 | 0/119 | 0/116 | 0/59
Major depression (Psychiatric disorders) | 0/119 | 1/118 | 0/119 | 0/119 | 0/116 | 0/59
Bladder prolapse (Renal and urinary disorders) | 0/119 | 0/118 | 0/119 | 0/119 | 1/116 | 0/59
Pelvic prolapse (Reproductive system and breast disorders) | 0/119 | 0/118 | 1/119 | 0/119 | 0/116 | 0/59
Uterine prolapse (Reproductive system and breast disorders) | 0/119 | 0/118 | 0/119 | 0/119 | 1/116 | 0/59
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0/119 | 0/118 | 1/119 | 0/119 | 0/116 | 0/59
Arterial hemorrhage (Vascular disorders) | 0/119 | 0/118 | 1/119 | 0/119 | 0/116 | 0/59
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | ABT-335 + 20 mg Simvastatin | ABT-335 + 40 mg Simvastatin | ABT-335 | 20 mg Simvastatin | 40 mg Simvastatin | 80 mg Simvastatin
Abdominal pain (Gastrointestinal disorders) | 1/119 | 4/118 | 3/119 | 1/119 | 1/116 | 0/59
Abdominal pain upper (Gastrointestinal disorders) | 4/119 | 2/118 | 3/119 | 1/119 | 2/116 | 2/59
Constipation (Gastrointestinal disorders) | 2/119 | 4/118 | 6/119 | 3/119 | 3/116 | 1/59
Diarrhea (Gastrointestinal disorders) | 2/119 | 5/118 | 5/119 | 5/119 | 9/116 | 4/59
Dyspepsia (General disorders) | 5/119 | 7/118 | 8/119 | 3/119 | 6/116 | 1/59
Nausea (Gastrointestinal disorders) | 3/119 | 5/118 | 5/119 | 4/119 | 5/116 | 1/59
Vomiting (Gastrointestinal disorders) | 0/119 | 2/118 | 2/119 | 1/119 | 1/116 | 2/59
Fatigue (General disorders) | 0/119 | 2/118 | 4/119 | 3/119 | 0/116 | 1/59
Pain (General disorders) | 5/119 | 1/118 | 6/119 | 1/119 | 4/116 | 0/59
Influenza (Infections and infestations) | 3/119 | 3/118 | 0/119 | 2/119 | 4/116 | 2/59
Nasopharyngitis (Infections and infestations) | 9/119 | 9/118 | 7/119 | 11/119 | 4/116 | 1/59
Sinusitis (Infections and infestations) | 3/119 | 6/118 | 3/119 | 0/119 | 3/116 | 0/59
Upper respiratory tract infection (Infections and infestations) | 2/119 | 8/118 | 7/119 | 6/119 | 11/116 | 3/59
Joint sprain (Injury, poisoning and procedural complications) | 0/119 | 0/118 | 0/119 | 0/119 | 0/116 | 2/59
Alanine aminotransferase increased (Investigations) | 5/119 | 2/118 | 1/119 | 0/119 | 0/116 | 0/59
Aspartate aminotransferase increased (Investigations) | 4/119 | 2/118 | 0/119 | 0/119 | 0/116 | 0/59
Blood creatine phosphokinase increased (Investigations) | 4/119 | 1/118 | 0/119 | 1/119 | 3/116 | 2/59
Arthralgia (Musculoskeletal and connective tissue disorders) | 7/119 | 7/118 | 3/119 | 8/119 | 6/116 | 2/59
Back pain (Musculoskeletal and connective tissue disorders) | 10/119 | 4/118 | 9/119 | 8/119 | 9/116 | 2/59
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1/119 | 5/118 | 2/119 | 3/119 | 8/116 | 1/59
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3/119 | 2/118 | 0/119 | 2/119 | 4/116 | 0/59
Myalgia (Musculoskeletal and connective tissue disorders) | 5/119 | 3/118 | 6/119 | 4/119 | 6/116 | 3/59
Neck pain (Musculoskeletal and connective tissue disorders) | 2/119 | 1/118 | 1/119 | 0/119 | 5/116 | 0/59
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6/119 | 3/118 | 6/119 | 6/119 | 6/116 | 1/59
Dizziness (Nervous system disorders) | 4/119 | 0/118 | 5/119 | 3/119 | 1/116 | 2/59
Headache (Nervous system disorders) | 11/119 | 25/118 | 18/119 | 14/119 | 24/116 | 5/59
Hypoesthesia (Nervous system disorders) | 0/119 | 0/118 | 3/119 | 1/119 | 2/116 | 2/59
Sinus headache (Nervous system disorders) | 2/119 | 2/118 | 5/119 | 1/119 | 4/116 | 0/59
Pollakiuria (Renal and urinary disorders) | 0/119 | 4/118 | 0/119 | 0/119 | 0/116 | 0/59
Cough (Respiratory, thoracic and mediastinal disorders) | 4/119 | 7/118 | 3/119 | 5/119 | 5/116 | 3/59
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4/119 | 0/118 | 2/119 | 0/119 | 0/116 | 0/59
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5/119 | 2/118 | 4/119 | 1/119 | 0/116 | 0/59
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 4/119 | 3/118 | 3/119 | 1/119 | 2/116 | 0/59
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 3/119 | 1/118 | 2/119 | 2/119 | 4/116 | 1/59
Hypertension (Vascular disorders) | 0/119 | 3/118 | 0/119 | 0/119 | 2/116 | 2/59

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Not to publish or present the results before the publication of the multi-center investigator paper, but in no event shall be so restricted after the expiration of twelve (12) months from completion of the studies at all sites. Any presentation or publication to be submitted to Sponsor (in draft of the same) for Sponsor review and comment.